CLINICAL TRIAL: NCT01601067
Title: Integrated Alcohol Disorder and PTSD Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NURA-011-11F
Record Dates: First submitted 2012-02-28; First posted 2012-05-17 (Estimated); Results first posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: PTSD; Alcoholism
Keywords: posttraumatic stress disorder; psychotherapy; alcoholism
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Integrated Prolonged Exposure Therapy (Experimental): Integrated Prolonged exposure Psychotherapy (I-PE; PE integrated with elements of Integrated Cognitive Behavioral Therapy for alcohol use disorder)
  Interventions: Behavioral: Integrated Prolonged Exposure Therapy
- Arm 2: Seeking Safety (Active Comparator): Seeking Safety
  Interventions: Behavioral: Seeking Safety

INTERVENTIONS:
Behavioral: Integrated Prolonged Exposure Therapy — Prolonged exposure (PE) therapy is an evidence based practice for the treatment of PTSD. Components of PE included education about PTSD and exposure to avoided reminders of trauma.
  Other Names: I-PE
  Arms: Arm 1: Integrated Prolonged Exposure Therapy
Behavioral: Seeking Safety — Seeking Safety (SS) teaching coping skills in behavioral, cognitive, and interpersonal domains so that people are able to make safe choices rather than drinking or PTSD-related behaviors such as avoidance.
  Other Names: SS
  Arms: Arm 2: Seeking Safety

SUMMARY:
Comorbidity of alcohol use disorder (AD) and posttraumatic stress disorder (PTSD) is common. Currently available treatments often do not lead to sustained recovery from these disorders, possibly because they typically do not include exposure therapy which is considered best practice treatments for PTSD. This study compares exposure-based integrated treatment to integrated coping skills psychotherapy (a well disseminated practice) for comorbid AD and PTSD with the hypothesis that exposure therapy will allow those with PTSD to better sustain PTSD symptom reduction and reduction in alcohol use. The aim of this grant is to change common treatment practices for comorbid AD and PTSD by increasing the availability of evidence-based PTSD treatment for those with AD.

DETAILED DESCRIPTION:
Objectives. Co-occurrence of alcohol use disorder (AD) and posttraumatic stress disorder (PTSD) is common. Research supports exposure therapy as the front line treatment for PTSD as this approach is most likely to lead to sustained recovery from the disorder. However, individuals with AD are generally not offered exposure therapies because of beliefs that exposure would lead to engagement in greater alcohol use and other dangerous behaviors. Most research and clinical treatment for comorbid AD and PTSD (AD/PTSD) have involved coping skills based therapies that have generally not shown sustained reductions in alcohol use and PTSD symptoms. A growing body of evidence suggests these individuals with AD/PTSD are able to handle and benefit from exposure. This proposed trial will compare an integrated exposure psychotherapy to an integrated coping skills psychotherapy for the treatment of AD/PTSD. In addition, mechanisms of change for Veterans with AD/PTSD in both treatment conditions, including therapy process variables, changes in negative affect, and sleep problems, will be explored. This project addresses a critical barrier in the field - the widely held belief that individuals with AD and PTSD cannot tolerate exposure therapy, although it is the best practice treatment for PTSD. The fundamental rationale is to improve the evidence base that informs how patients with AD/PTSD can attain sustained recovery. The investigators propose a randomized controlled trial to evaluate an integrated exposure-based treatment for concurrent AD and PTSD. The primary aim will be to conduct a randomized controlled trial to evaluate the effects of integrated exposure psychotherapy when compared to a present-focused coping skills based intervention (Seeking Safety; SS) in 148 male and female Veterans who have AD and PTSD. The hypotheses are that at post-treatment both groups will show reductions in alcohol use, but the integrated exposure group will demonstrate greater reductions in PTSD symptoms than SS. At 5- and 8-month post-baseline follow-up, the integrated exposure group will have significantly fewer percent drinking days and fewer PTSD symptoms than SS. In addition, mechanisms of change in both treatment conditions will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Veterans who were victims of psychological trauma that occurred in childhood or adulthood.
* At least one month post-trauma.
* Age 18 or older.
* Meeting diagnostic criteria for current alcohol dependence and PTSD.
* Literate in English.
* Intend to stay in San Diego during study participation.
* Willing to attend psychotherapy and measurement sessions.
* Willing to stay cut down alcohol use significantly during treatment.

Exclusion Criteria:

* Moderate or severe cognitive impairment on the Brief Neuropsychological (NP) Assessment Battery as this may interfere with ability to benefit from treatment.
* Acutely suicidal individuals will be referred for more appropriate treatment.
* Histories of psychosis or mania independent of substance use will be excluded because the presence of these disorders can impede therapy progress.
* Individuals who use intravenous drugs will be excluded.
* Participants who do not have adequate memory of the trauma will be excluded because such memory is necessary for exposure therapy.
* Only Veterans residing within 50 miles of the site will be included.
* Those with life threatening or unstable medical illness, documented neurological disorder, or inability to read will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2013-01-21 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonya B. Norman, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Not in our approval.

REFERENCES:
- [Derived] Lyons R, Helm J, Luciano M, Haller M, Norman SB. The role of posttraumatic cognitions in integrated treatments for co-occurring posttraumatic stress disorder and alcohol use disorder. Psychol Trauma. 2024 Dec;16(Suppl 3):S532-S539. doi: 10.1037/tra0001540. Epub 2023 Jun 29. PMID 37384482
- [Derived] Marx BP, Lee DJ, Norman SB, Bovin MJ, Sloan DM, Weathers FW, Keane TM, Schnurr PP. Reliable and clinically significant change in the clinician-administered PTSD Scale for DSM-5 and PTSD Checklist for DSM-5 among male veterans. Psychol Assess. 2022 Feb;34(2):197-203. doi: 10.1037/pas0001098. Epub 2021 Dec 23. PMID 34941354
- [Derived] Tripp JC, Haller M, Trim RS, Straus E, Bryan CJ, Davis BC, Lyons R, Hamblen JL, Norman SB. Does exposure exacerbate symptoms in veterans with PTSD and alcohol use disorder? Psychol Trauma. 2021 Nov;13(8):920-928. doi: 10.1037/tra0000634. Epub 2020 Jul 16. PMID 32673006
- [Derived] Tripp JC, Angkaw A, Schnurr PP, Trim RS, Haller M, Davis BC, Norman SB. Residual Symptoms of Posttraumatic Stress Disorder and Alcohol Use Disorder Following Integrated Exposure Treatment Versus Coping Skills Treatment. J Trauma Stress. 2020 Aug;33(4):477-487. doi: 10.1002/jts.22552. Epub 2020 Jun 18. PMID 32557843
- [Derived] Capone C, Tripp JC, Trim RS, Davis BC, Haller M, Norman SB. Comparing Exposure- and Coping Skills-Based Treatments on Trauma-Related Guilt in Veterans With Co-Occurring Alcohol Use and Posttraumatic Stress Disorders. J Trauma Stress. 2020 Aug;33(4):603-609. doi: 10.1002/jts.22538. Epub 2020 Jun 10. PMID 32521096
- [Derived] Norman SB, Trim R, Haller M, Davis BC, Myers US, Colvonen PJ, Blanes E, Lyons R, Siegel EY, Angkaw AC, Norman GJ, Mayes T. Efficacy of Integrated Exposure Therapy vs Integrated Coping Skills Therapy for Comorbid Posttraumatic Stress Disorder and Alcohol Use Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2019 Aug 1;76(8):791-799. doi: 10.1001/jamapsychiatry.2019.0638. PMID 31017639

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants contacted our study in response to 1) flyers posted in VA mental health, primary care, and alcohol and substance use treatment programs; 2) from advertisements in print and web-based media; and 3) by VA primary care, SAMI, PTSD, and other psychiatry clinics
Pre-assignment Details: Enrolled participants were excluded from the study for the following reasons: 27 did not meet inclusion criteria; 15 did not complete intake or did not return for intake following informed consent;5 refused research after consent; 2 had travel or logistical constrains.
Period: Overall Study
Arm/Group | Arm 1: Integrated Prolonged Exposure Therapy | Arm 2: Seeking Safety
Started | 63 | 56
Completed | 30 | 34
Not Completed | 33 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Integrated Prolonged Exposure Therapy | Arm 2: Seeking Safety | Total
Number analyzed (Participants) | 63 | 56 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (13.5) | 39.7 (11.3) | 41.6 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 56 | 51 | 107
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 41 | 37 | 78
  Black | 8 | 8 | 16
  Asian | 3 | 3 | 6
  Other | 11 | 7 | 18
  Unavailable | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 63 | 56 | 119

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale (CAPS)
Description: The CAPS-5 (score range, 0-80, with 0 indicating no PTSD symptoms and 80 indicating extreme ratings across all symptoms), a 30-item structured interview considered to be the criterion standard for PTSD, was the primary measure of PTSD symptoms and diagnosis. Diagnosis was determined using the rule of a severity score of 2 or higher, which follows DSM-5 PTSD criteria.
Time Frame: baseline through 6 month follow-up
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1: Integrated Prolonged Exposure Therapy | Arm 2: Seeking Safety
Number analyzed (Participants) | 63 | 56
score on a scale
  Baseline | 43.2 [40.0 to 46.4] | 42.1 [38.7 to 45.5]
  After Treatment | 25.8 [22.1 to 29.6] | 32.9 [29.3 to 36.6]
  3 month follow-up | 26.4 [22.6 to 30.3] | 31.0 [27.0 to 35.1]
  6 month follow-up | 22.5 [18.2 to 26.8] | 29.8 [25.6 to 33.9]
Statistical Analysis 1: Comparison: Arm 1: Integrated Prolonged Exposure Therapy vs Arm 2: Seeking Safety; Test type: Superiority; p = .002, Mixed Models Analysis

2. Secondary Outcome: Timeline Follow-Back Procedure (TLFB) for Alcohol Use
Description: Frequency and quantity of alcohol use were assessed using the Timeline Follow-Back, a calendar-assisted structured clinical interview that displays good psychometric properties. The PHDD was calculated by dividing the number of days in which 5 or more drinks for men or 4 or more drinks for women were consumed by the total number of days in the reference period.
Time Frame: baseline to 6-month follow-up
Measure: Mean (95% Confidence Interval); unit: percentage of days
Arm/Group | Arm 1: Integrated Prolonged Exposure Therapy | Arm 2: Seeking Safety
Number analyzed (Participants) | 63 | 56
percentage of days
  % Days heavy drinking - baseline | 52.5 [46.5 to 58.6] | 50.4 [44.1 to 56.7]
  % Days heavy drinking -After treatment | 21.0 [13.4 to 28.6] | 17.4 [10.4 to 24.5]
  % Days heavy drinking - 3 month follow up | 14.2 [6.9 to 21.4] | 15.0 [7.1 to 22.8]
  % Days heavy drinking - 6-month follow-up | 20.2 [11.9 to 28.5] | 19.9 [12.1 to 27.6]
  % Days abstinent - baseline | 34.3 [27.1 to 41.6] | 31.2 [23.5 to 38.8]
  % Days abstinent - After treatment | 67.5 [58.9 to 76.1] | 63.1 [54.9 to 71.4]
  % Days abstinent - 3-month follow up | 65.6 [57.0 to 74.2] | 68.4 [59.3 to 77.4]
  % Days abstinent - 6-month follow-up | 66.2 [56.5 to 75.9] | 64.0 [54.8 to 73.3]
Statistical Analysis 1: Comparison: Arm 1: Integrated Prolonged Exposure Therapy vs Arm 2: Seeking Safety; Test type: Superiority; p = .91, Mixed Models Analysis — heavy drinking days

ADVERSE EVENTS:
Time Frame: Four years and seven months
Arm/Group | Arm 1: Integrated Prolonged Exposure Therapy | Arm 2: Seeking Safety
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/56
Serious Adverse Events (participants affected / at risk) | 2/63 | 0/56
Other Adverse Events (participants affected / at risk) | 0/63 | 0/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Integrated Prolonged Exposure Therapy (N=63) | Arm 2: Seeking Safety (N=56)
hospitalization for alcohol intoxication and mood stabilization (Psychiatric disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
- Mostly male veteran sample

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-04-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT01601067/Prot_000.pdf
  • Statistical Analysis Plan (2011-09-03): https://cdn.clinicaltrials.gov/large-docs/67/NCT01601067/SAP_001.pdf